CLINICAL TRIAL: NCT01071512
Title: Tysabri Effects on Cognition and Neurodegeneration in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-094A
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Multiple Sclerosis
Keywords: MRI; OCT; Tysabri; Multiple Sclerosis; cognition
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tysabri (Experimental): Natalizumab 300 mg IV every 4 weeks
  Interventions: Drug: Tysabri

INTERVENTIONS:
Drug: Tysabri — Infuse TYSABRI® 300 mg in 100 mL 0.9% Sodium Chloride Injection, USP over approximately one hour. After the infusion is complete, flush with 0.9% Sodium Chloride Injection, USP. Tysabri will be infused every four weeks.
  Other Names: Natalizumab

SUMMARY:
The long-term objective is to further establish the role of Tysabri in preventing neurological degeneration in multiple sclerosis (MS) and to establish powerful and efficient new markers for neurological degeneration in MS. The study intends to correlate cognition with two instruments and their measurements-MRI and OCT (optical coherence tomography).

DETAILED DESCRIPTION:
The specific aims are:

1. To determine the effects of Tysabri on cognition (memory, thought processes, etc.)
2. To determine the effects of Tysabri on specific MRI markers for cognitive dysfunction
3. To determine the effects of Tysabri on retinal nerve fiber layer thickness (RNFL) using optical coherence tomography (OCT), a special instrument used in ophthalmology

ELIGIBILITY:
Inclusion Criteria:

* 18 through 60 years of age inclusive
* Diagnosis of relapsing remitting multiple sclerosis
* Prior to treatment phase, have had disease activity with at least 1 documented relapse during the previous year OR 2 documented relapses during the previous 2 years OR one or more new MRI lesions (Gd+ and/or T2 hyperintense)
* An Expanded Disability Status Scale (EDSS) score of 0-4.5 inclusive
* Neurologically stable with no evidence of relapse or corticosteroid treatment within 30 days prior to treatment
* Never been treated with Tysabri/natalizumab.

Exclusion Criteria:

* Another type of MS other than relapsing remitting multiple sclerosis (RRMS)
* A history of chronic disease of the immune system other than MS or a known immunodeficiency syndrome/immunocompromised
* A history or presence of cancer (except for successfully treated basal or squamous cell carcinoma of skin)
* Active systemic bacterial, viral or fungal infections, or diagnosis of AIDS, Hepatitis B, Hepatitis C infection defined as a positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests, respectively
* Have received any live or live attenuated vaccines (including for varicella-zoster virus or Measles) within the last 2 months
* Have received total lymphoid irradiation or bone marrow transplantation
* Have been treated with: corticosteroids or adrenocorticotropic hormones (ACTH) within the last month, IFN-β or glatiramer acetate within the last 3 months, immunosuppressive medications such as azathioprine or methotrexate within the last 6 months, immunoglobulins and/or monoclonal antibodies (including natalizumab) within the last 6 months, or cladribine, cyclophosphamide or mitoxantrone at any time.
* Any medically unstable condition or a progressive neurological disorder, other than MS, which may affect participation in the study
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal or other major disease
* Unable to undergo MRI scans, including claustrophobia, have a pacemaker or history of hypersensitivity to gadolinium-DTPA
* Have had a relapse within 30 days prior AND/OR not stabilized from a previous relapse
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity to natalizumab/Tysabri
* A clinically significant infectious disease, such as cellulitis, pneumonia, septicemia
* History of progressive multifocal leukoencephalopathy(PML)
* Participation in any clinical research study evaluating another investigational drug or therapy within the last 6 months
* History of Tysabri therapy
* Abnormal screening blood test
* Females who are not postmenopausal for at least 1 year, surgically sterile or willing to practice effective contraception during the study
* Nursing mothers, pregnant women, and women planning to become pregnant while on study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Bernard, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tysabri
Started | 20
Completed | 15
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Development of antibodies to drug | 2
Not completed — positive anti-JC virus antibody test | 2

BASELINE CHARACTERISTICS:
Population: Includes patients that completed treatment
Arm/Group | Tysabri
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8
  African-American | 6
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function Over Time
Description: Cognitive function was assessed using the oral version of the Symbol Digit Modalities Test (SDMT). The number of correct responses in 90 seconds was recorded (possible range 0-110). For analysis, SDMT scores were converted to z-scores using published age and education based norms. A negative z-score indicates a SDMT score below the mean based on the age and education based norms, for example a z-score of -2 = 2 standard deviations below the mean; a positive z-score indicating a score above the mean. Higher scores indicate better cognitive function.
Time Frame: Baseline, 48 weeks, 96 weeks
Population: Summary statistics are based on the 15 subjects who completed treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tysabri
Number analyzed (Participants) | 15
units on a scale
  Baseline | -1.5 (0.9)
  Week 48 | -1.2 (1.0)
  Week 96 | -1.2 (0.9)
Statistical Analysis 1: Comparison: Tysabri; Analysis used all available data from subjects, including those who dropped out early; Test type: Other; p = 0.17, Mixed Models Analysis

2. Secondary Outcome: Change Over Time in Retinal Nerve Fiber Layer Thickness
Description: Retinal Nerve Fiber Layer (RNFL) thickness was measured using spectral domain OCT scans by a trained technician. Scans were performed without pupil dilation.
Time Frame: Baseline, 24, 48, 72, and 96 weeks
Population: Summary statistics are provided based on subjects completing all treatment
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Tysabri
Number analyzed (Participants) | 15
micrometer
  Baseline | 86 (13)
  Week 24 | 85 (12)
  Week 48 | 85 (13)
  Week 72 | 85 (13)
  Week 96 | 85 (13)
Statistical Analysis 1: Comparison: Tysabri; Analysis used all available data; Test type: Other; p = 0.6, Mixed Models Analysis

3. Secondary Outcome: Change Over Time in Brain Parenchymal Fraction
Description: Measured based on MRI scan on a 3T Phillips scanner. This is a measure of brain atrophy (i.e., brain volume loss) with lower values indicating greater atrophy (possible range 0-1).
Time Frame: Baseline, 48 weeks, 96 weeks
Population: Summary statistics are based on subjects completing treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tysabri
Number analyzed (Participants) | 15
units on a scale
  Baseline | 0.970 (0.011)
  Week 48 | 0.969 (0.012)
  Week 96 | 0.971 (0.014)
Statistical Analysis 1: Comparison: Tysabri; Analysis used all available data; Test type: Other; p = 0.3, Mixed Models Analysis

4. Secondary Outcome: Change Over Time in Normalized Thalamic Volume
Description: Measured on MRI scan
Time Frame: Baseline, 48 weeks, 96 weeks
Population: Summary statistics are based on subjects completing all treatment
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tysabri
Number analyzed (Participants) | 15
mL
  Baseline | 13.9 (1.9)
  Week 48 | 13.7 (2.0)
  Week 96 | 13.7 (2.1)
Statistical Analysis 1: Comparison: Tysabri; Analysis used all available data; Test type: Other; p = 0.02, Mixed Models Analysis

5. Secondary Outcome: Change Over Time in Normalized Hippocampal Volume
Description: Measured on MRI scan
Time Frame: Baseline, 48 weeks, 96 weeks
Population: Summary statistics are based on subjects completing all treatment
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tysabri
Number analyzed (Participants) | 15
mL
  Baseline | 6.8 (0.8)
  Week 48 | 6.7 (1.0)
  Week 96 | 6.6 (0.9)
Statistical Analysis 1: Comparison: Tysabri; Analysis used all available data; Test type: Other; p = 0.9, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 96 weeks
Arm/Group | Tysabri
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tysabri (N=20)
pruritis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes